CLINICAL TRIAL: NCT03364374
Title: Biomechanical Assessment of the Relationship Between Postural Control and Fine Motor Skills in People With Stroke
Brief Title: Postural Control and Fine Motor Skills in People With Stroke
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christian Finetto, Post-doctoral Scholar, Medical University of South Carolina
Other Study IDs: Pro00040824
Record Dates: First submitted 2017-11-27; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Upper extremity; Posture
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke survivors: Individuals that experienced uni-hemispheric ischemic or hemorrhagic stroke
  Interventions: Behavioral: Postural counseling
- Controls: Healthy controls with no history of stroke
  Interventions: Behavioral: Postural counseling

INTERVENTIONS:
Behavioral: Postural counseling — A therapist will provide verbal/physical cues to improve the participants posture

SUMMARY:
This study evaluates the relationship between seated posture and fine motor performance in a drawing task in people with stroke and in healthy control subjects.

DETAILED DESCRIPTION:
Current stroke rehabilitation practice guidelines support an interprofessional approach which integrates discipline-specific goals into a comprehensive plan of care. However, there has been a failure to implement interprofessional guidelines into today's stroke rehabilitation clinical practice. Instead it is common that one discipline focuses on recovery of posture, while another discipline focuses on recovery of fine motor skills. The investigators argue that control of the hand is not independent from postural control. In fact, treating them separately ignores the kinematic and muscular linkages connecting the trunk to the hand via the scapula and proximal arm. It also ignores evidence that postural and hand muscles have overlapping cortical representations thus likely have similar neural control networks. Hence, the overall goal of this project is to demonstrate the relationship of posture and fine motor skills to advance stroke rehabilitation.

The study will include two groups, stroke survivors and neurologically healthy controls, and both will perform a tracing task while seated on a backless bench. The task will be performed twice, at baseline and after giving participants cues to improve their posture. Both task repetitions will be performed in a single session on the same day. Kinetic and kinematic data will be collected to evaluate posture, postural stability and fine motor performance. Data collected at baseline will be used to examine the relationship between postural impairments and fine motor deficits. Additionally, we will evaluate the effects of postural cues on body segment alignment, stability and fine motor performance.

ELIGIBILITY:
Stroke survivors:

Inclusion Criteria:

* experienced uni-hemispheric ischemic or hemorrhagic stroke 3 mo - 7 yrs prior
* ability to grasp and hold a stylus for the duration of the experiments
* passive motion throughout the paretic UE within 20° of normal
* dominant side affected

Exclusion Criteria:

* lesion in brainstem or cerebellum
* presence of other neuro-disease impairing motor skills
* unable to understand 3-step directions
* pain, orthopedic condition or impaired corrected vision that would alter reaching

Healthy Controls:

Inclusion Criteria:

* no history of stroke or incomplete spinal cord injury
* no medical, orthopedic, neurological, or uncorrected visual condition that would limit the ability to participate in upper extremity testing

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients will be recruited from the MUSC Center for Rehabilitation Research in Neurological Conditions database (approved IRB PRO# 15991, PI Kautz) that currently contains contact information for ~120 stroke survivors who have agreed to be contacted for research participation.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Change in tracing smoothness from baseline to after postural counseling | Within 24 hours
  Change in the average jerk of the hand trajectory during a tracing task

SECONDARY OUTCOMES:
Change in center of pressure displacement from baseline to after postural counseling | Within 24 hours
  Change in the maximum center of pressure displacement during a tracing task

CONTACTS AND LOCATIONS:
Overall Officials: Christian Finetto, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided